CLINICAL TRIAL: NCT05092399
Title: Differential Effects of Very Low-Calorie Diet (VLCD), Roux-En-Y-Gastric Bypass and Sleeve Gastrectomy on Pancreatic, Liver, Muscle and Heart Fat Deposition and Metabolism in People With Type 2 Diabetes: An MRI Study
Brief Title: Effects of VLCD and Bariatric Surgery in Patients With Type 2 Diabetes
Acronym: BARIATRICMRI
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: University of Leicester (Other); Medical Research Council (Other Government); International Stem Cell Forum (Other); University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 21047
Record Dates: First submitted 2021-09-06; First posted 2021-10-25 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2023-11

CONDITIONS: Type2 Diabetes; NAFLD; Obesity
Keywords: VLCD; Bariatric Surgery; MRI; MRS
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RYGB: Patients undergoing Roux-en-Y gastric bypass surgery
  Interventions: Procedure: Bariatric Surgery
- SG: Patients undergoing Sleeve Gastrecomy surgery
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — No study interventions

SUMMARY:
The investigators are therefore interested to explore the effects of VLCD and different bariatric surgery procedures to changes in the physical deposition of fat in organs which regulate glucose metabolism (i.e. in the liver, pancreas, muscle) in the earlier (6 weeks) and intermediate (4 months) period after bariatric surgery, where rate of weight loss at this stage are similar between the two procedures. Increased understanding of the changes in these important metabolic organs, will increase the investigators' understanding of mechanism of diabetes remission following bariatric surgery, their effects on weight loss or changes in gut hormones levels. Magnetic Resonance imaging (MRI) and Magnetic Resonance spectroscopy (MRS) are non-invasive, non-ionising techniques. MRI can be used to investigate the body's physiology and MRS can be used to investigate the body's metabolic processes, so by combining these two methods the investigators are able to investigate the process of fat reduction and diabetes remission post gastric surgery without performing any secondary invasive procedures The purpose of this project is to investigate the effects of a Very Low Calorie Diet (VLCD) followed by two different bariatric surgical procedures, Roux-en-Y Gastric Bypass (RYGB) and Sleeve gastrectomy (SG) on skeletal muscle, liver and pancreatic fat deposition, ATP flux as well as cardiac function.

DETAILED DESCRIPTION:
There are NO research interventions, this study is observing a patient's response to clinical interventions. The below describes the investigators methods of observation.

Screening:

Participants who are listed for surgery by the Bariatric surgical Tier 4 MDT team will be approached by one of the main care team who may also be a member of the research team during the ERAS session (Enhanced Recovery After Surgery) approximately 6 months before surgery. If the participants wish to partake in the study the will be then screened for ability and willingness to undergo MRI in order to prevent any wasting of the patients time and prevent unnecessary data storage. If eligible and consent is provided, their details will be kept by the research team to be contacted for further appointment to attend the investigators University of Nottingham (UoN) research unit based at the Royal Derby Hospital.

There are 2 main arms to the study, consists of 2 arms, patients undergoing RYGB (group 1) and Patients undergoing SG (group 2) Within these groups there are category A and B participants.

Category A - Primary Study - Participants who will be used to investigate the primary and secondary outcomes.

Category B - Exploratory sub-study - Participants will be used to investigate the Primary outcome but also as a pilot set of data for cardiac measures.

At all category A sessions Participants will be asked to attend a session at the Sir Peter Mansfield Imaging Centre (SPMIC) on the UoN main campus.

The participants will receive an MRI and MRS scan, a Blood Test and a liquid mixed meal test at every session. The mixed meal test is not apart of routine care, in this study it shall be used to examine the change in participants response to a meal after each clinical intervention (VLCD and Surgery). Blood samples will be taken by a trained member of staff and transferred to the Royal Derby Hospital for testing, this is to obtain Glucose, Ghrelin, C-peptide, glucagon and total and intact glucagon-like peptide-1 (GLP-1).

Participants in category B will be asked to attend sessions at the SPMIC. And will only receive MRI and MRS scans.

Session 1:

A member of the research team will reach out to the patient 2 weeks prior to the commencement of their VLCD in order to confirm the participants are still interested in participating, book in the first study session and answer any questions the participants may have.

Session 2:

Between 3 and 1 day prior to the commencement of the VLCD.

Category A:

The MRI protocol for this session physiology scans of the Chest, Abdomen and Skeletal Muscle (thigh) and MRS is proton spectroscopy performed on the Liver. Participants will be in the scanner for no longer than 1 hour.

Category B:

Basic Cardiac measures using MRI will be used in planning for Proton and Phosphorus MR Spectroscopy (MRS). Participants will be offered a break after being in the scanner for 1hour with a maximum time in the scanner of 2hours.

Session 3:

Between 3 and 1 day prior to the Participants Bariatric Surgery.

Category A:

The MRI protocol for this session is physiology scans for the Chest, Abdomen and Skeletal Muscle (thigh) and MRS is proton spectroscopy and a 31P (phosphorous) spectroscopy performed on the Liver. Basic. Participants will be offered a break after being in the scanner for 1hour with a maximum time in the scanner of 2hours.

Category B:

Basic Cardiac measures using MRI will be used in planning for Proton and Phosphorus MR Spectroscopy (MRS). Participants will be offered a break after being in the scanner for 1hour with a maximum time in the scanner of 2hours

Surgery:

Roux-en-Y Gastric Bypass (RYGB): Follows standard clinical practice. Sleeve Gastrectomy (SG): Follows standard clinical practice.

Session 4:

6 weeks post Bariatric Surgery.

Category A:

The MRI protocol for this session is physiology scans of the Chest, Abdomen and Skeletal Muscle (thigh) and MRS is proton spectroscopy and a 31P (phosphorous) spectroscopy performed on the Liver. Participants will be offered a break after being in the scanner for 1hour with a maximum time in the scanner of 2hours.

Category B:

Basic Cardiac measures using MRI will be used in planning for Proton MR Spectroscopy (MRS). Participants will be in the scanner for no longer than 1 hour.

Session 5:

16 weeks post Bariatric Surgery.

Category A:

The MRI protocol for this session is physiology scans of the Chest, Abdomen and Skeletal Muscle (thigh) and MRS is proton spectroscopy on the Liver. Participants will be in the scanner for no longer than 1 hour.

Category B:

Basic Cardiac measures using MRI will be used in planning for Proton MR Spectroscopy (MRS). Participants will be in the scanner for no longer than 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Listed for RYCG or SG at the royal derby hospital
* BMI>/=18
* Type 2 diabetes
* Ability to give informed consent

Exclusion Criteria:

1. If they are not suitable for either RYGB or SG as determined by the MDT meeting
2. BMI>60
3. Liver cirrhosis.
4. Participants will be excluded if they are deemed unfit for an MRI via the standard safety screening form.
5. Participants will be excluded if their waist circumference is too large for them to safely fit inside the bore of the MRI with surface coils added.
6. Participation in other research projects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living in and around Derby and Leicester who are attending the bariatric clinic at royal derby hospital.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Effects of VLCD | baseline to +2weeks
  Changes to liver fat volume due to VLCD as measured with MRI

SECONDARY OUTCOMES:
Effects of VLCD on Liver and Pancreas | baseline to +2weeks
  Changes to live and pancreatic fat as measured using MRI and MRS as measured as percentage fat in tissue.
Effects of VLCD and bariatric surgery | +2weeks to +6weeks(post surgery)
  Changes to Skeletal muscle liver and pancreatic fat as measured using MRI and MRS as measured as percentage fat in tissue.
Effects of VLCD and bariatric surgery | +6weeks(post surgery) to +4months (post surgery)
  Changes to Skeletal muscle, liver and pancreatic fat as measured using MRI and MRS as measured as percentage fat in tissue
Effects of VLCD and bariatric surgery | +2weeks to +6weeks (post surgery)
  Changes to Liver ATP flux as measured using MRS
Effects of VLCD and bariatric surgery | +6weeks (post surgery) to +4months (post surgery)
  Changes to Liver ATP flux as measured using MRS
Difference between surgery types (RYGB Vs SG) | +6weeks (post surgery)
  Changes to Liver ATP flux as measured using MRS
Effects of different surgery types (RYGB Vs SG) on Liver ATP flux | +4months (post surgery)
  Changes to Liver ATP flux as measured using MRS
Effects of different surgery types (RYGB Vs SG) on Organ fat content | +4months (post surgery)
  Changes to skeletal muscle, liver and pancreatic fat as measured using MRI and MRS as measured as percentage fat content of tissue
Difference between surgery types (RYGB Vs SG) | +6 weeks (post surgery)
  Changes to Skeletal muscle, liver and pancreatic fat as measured using MRI and MRS as measured as percentage fat content of tissue
Effects of VLCD and bariatric surgery | 0 to +2weeks
  Bile Acid Quantification
Effects of VLCD and bariatric surgery | +6weeks post surgery
  Bile Acid Quantification
Effects of VLCD and bariatric surgery | 4months post surgery
  Bile Acid Quantification

CONTACTS AND LOCATIONS:
Overall Officials: Penny Gowland, Principal Investigator — University of Nottingham
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No